CLINICAL TRIAL: NCT01281683
Title: Dynamic Contrast-enhanced Magnetic Resonance Imaging in Evaluation of Liver Functional Status and Treatment Efficacy in Patients With Hepatocellular Carcinoma After Locoregional Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Tiffany Ting-Fang Shih, National Taiwan University Hospital
Other Study IDs: 201010059R
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TACE
- RFA

SUMMARY:
Hepatocellular carcinoma (HCC) is a major health problem worldwide. For patients with intermediate-stage disease, i.e., large or multifocal HCC without vascular invasion or extrahepatic spread, transarterial chemoembolization (TACE) is recommended as first line therapy with survival advantages. TACE can be performed repeatedly in patients with recurrent tumors who have adequate liver function reserves.

Two clinical issues of TACE remain un-resolved. The first issue is the possibility of TACE-induced liver parenchymal damage, which may influence further treatment options and outcome of the patients. Conventional ways to evaluate liver functional reserves, including Child-Pugh score, biochemistry and metabolic tests, and ultrasound elastography, are relatively non-specific. The second issue is the difficulty in evaluating TACE efficacy, which cannot be reliably measured by conventional, volumetric response criteria. Both issues should be resolved to optimize patient care.

Recently dynamic contrast-enhancing magnetic resonance imaging (DCE-MRI) is increasingly used to analysis perfusion changes of the liver, and can be applied to both liver parenchyma and tumors. Previous studies have shown clinical applications of perfusion imaging, such as evaluating the severity of liver fibrosis and cirrhosis, assessing the effectiveness of anti-angiogenic therapy, and evaluating tumor viability after locoregional therapy. DCE-MRI can be performed with a hepatobiliary specific contrast agent, Gd-EOB-DTPA (Gadoxetic acid, Primovist®, Bayer Schering), with dual benefit of dynamic phase and the delayed hepatobiliary phase imaging. The hepatobiliary phase imaging can provide additional information for hepatic lesion characterization and the functional status of the hepatocytes. We hypothesize that imaging parameters of DCE-MRI with Gd-EOB-DTPA could reflect non-tumorous liver parenchymal changes and can be used to predict and monitor treatment response in patients with HCC after TACE.

In this prospective cohort study, we will recruit patients referred for TACE with newly-diagnosed unresectable HCC or tumor recurrence after operation. Patients treated with radiofrequency ablation (RFA) will be recruited as a control group, since RFA is associated with minimal damage to the non-tumorous liver parenchyma. Key eligible criteria include chronic hepatitis B, histological or clinical diagnosis of HCC, tumors that are not amenable to surgical treatment and referred for TACE or RFA, ECOG performance status 0 or 1, Child-Pugh class A or B liver function, and measurable tumors (by RECIST 1.1). Eligible patients will receive the designated treatment (TACE or RFA) according to the current HCC treatment guidelines. DCE-MRI with Gd-EOB-DTPA will be used to analyze the non-tumorous liver parenchymal changes and treatment response, and will be performed at baseline, 3 days and 1 month after treatment, and then every 3 months for a maximum of 2 years. The primary endpoint of this study is progression of liver function reserve. The estimated time for patient recruitment is about half a year, and 40 patients and 20 patients will be recruited in the TACE and the RFA treatment group, respectively. The imaging parameters of the non-tumorous parenchyma and the tumors will be analyzed and correlated with clinical liver function parameters, and hepatic functional and tumor outcome of the patients.

ELIGIBILITY:
Inclusion Criteria:

6.1.1. HCC diagnosed according to the AASLD guideline1: tumor size > 1cm in a cirrhotic liver with typical appearance in one dynamic imaging study (hypervascular in the arterial phase with washout in the portal venous or delayed phase), or the tumor is biopsied.

6.1.2. Patients who had undergone surgery for the treatment of HCC are allowed. 6.1.3. At least one measurable tumor, according to RECIST version 1.1. 6.1.4. Age 18 years. 6.1.5. Chronic hepatitis B. 6.1.6. ECOG performance status 0 or 1. 6.1.7. Life expectancy 2 months. 6.1.8. Child-Pugh class A or B liver function with a Child-Pugh score of ≦ 8. 6.1.9. Liver transaminases (ALT and AST) 300 IU/L; total bilirubin 2 mg/dL; serum creatinine 2 mg/dL.

6.1.10.Specific criteria for the TACE cohort: tumors distributed within one lobe and with maximal diameter of 10cm (for adequate amount of non-tumorous liver parenchyma for evaluation).

6.1.11.Specific criteria for the RFA cohort: single tumor with size of less than 5cm in diameter or tumors 3 or less in number with size of less than 3cm in diameter. The target tumor(s) can be approached by ultrasound guidance.

Exclusion Criteria:

6.2.1. Chronic hepatitis C. 6.2.2. Diffuse or infiltrative pattern of disease. 6.2.3. Previous TACE procedure for treatment of HCC. 6.2.4. Hepatic artery, hepatic vein, or portal venous thrombosis. 6.2.5. History of HCC tumor rupture. 6.2.6. Presence of extra-hepatic metastases. 6.2.7. Documentation of large intrahepatic or portal-caval shunts. 6.2.8. Contraindication for DCE-MRI, including known contrast allergy, electronically operated implants or devices, and claustrophobia.

6.2.9. Unable to cooperate well with breath holding comments during MRI examination or RFA treatment.

6.2.10.Major systemic diseases that the investigator considers inappropriate for participation.

6.2.11.Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation and in the judgment of the investigator would make the patient inappropriate for entry into this study.

6.2.12.Coagulation abnormality, including platelet count < 50000/L, prolongation of prothrombin time 5 seconds or INR >1.5) which could not be corrected by component therapy.

6.2.13.Obvious ascites which possibly cause bleeding complication. 6.2.14.History or clinically significant cardiac arrhythmia that is considered risky for invasive procedures including TACE or RFA.

6.2.15.Woman who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for TACE or RFA with newly-diagnosed unresectable HCC or tumor recurrence after operation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-01

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Ting-Fang Shih, MD, Principal Investigator — Department of Medical Imaging, National Taiwan University Hospital.
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan